CLINICAL TRIAL: NCT00069238
Title: Phase 2 Trial of Alemtuzumab and Dose-Adjusted Epoch in Chemotherapy Naive Aggressive T and NK-Cell Lymphomas
Brief Title: Campath-1H and EPOCH to Treat Non-Hodgkin's T- and NK-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030304; 03-C-0304; NCT00072254 (obsolete NCT alias)
Record Dates: First submitted 2003-09-17; First posted 2003-09-18 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell
Keywords: Lymphoma; T-Cell Lymphoma; NK -Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell; Lymphoma | interventions — Alemtuzumab; Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alemtuzumab Dose Escalation (Experimental): Alemtuzumab (Campath) followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) every 3 weeks for up to 6 cycles. Three cohorts of 3 to 6 patients will be treated. Cohort 1 will receive 30mg of Alemtuzumab, cohort 2 will receive 60mg of Alemtuzumab, and cohort 3 will receive 90mg of Alemtuzumab. If 1 of 3 participants entered at a given dose level experiences dose limiting toxicity (DLT), up to 3 additional participants will be entered at that dose level. If 2 of 6 participants experience DLT at a particular dose level, the maximum tolerated dose (MTD) has been exceeded. The preceding dose level will be the MTD, provided 6 participants have been entered at this level and no more than 1 has experienced DLT.
  Interventions: Biological: Alemtuzumab (Campath); Drug: EPOCH

INTERVENTIONS:
Biological: Alemtuzumab (Campath) — Alemtuzumab (Campath) followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) every 3 weeks for up to 6 cycles.
  Other Names: Campath
Drug: EPOCH — Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) + Alemtuzumab (Campath) every 3 weeks for up to 6 cycles.
  Other Names: Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin

SUMMARY:
Background:

The paradigm of combining therapeutic agents with non-overlapping toxicities for the treatment of malignancy produces clinical remissions and cures in a number of tumor types.

A new class of agents, humanized and chimerized monoclonal antibodies, typically have little or no hematopoietic toxicity and can be readily combined with full doses of cytotoxic chemotherapy. It has become clear that in certain lymphomas and breast cancers, the combination of monoclonal antibodies and chemotherapy improves response rate and the quality of the response compared with that achieved by treatment with either agent alone.

The clinical outcome for patients with T-cell non-Hodgkins lymphoma is significantly inferior to the outcome of patients with B-cell non-Hodgkin s lymphoma. In most reports less than 20% of patients with T cell lymphoid malignancies remain free of disease at 5 years.

Objectives:

Determine the toxicity of Alemtuzumab and etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) chemotherapy in untreated cluster of differentiation 52 (CD52)-expressing T and natural killer (NK) lymphoid malignancies.

Determine the maximum tolerated dose of Alemtuzumab administered in combination with EPOCH chemotherapy.

Determine in a preliminary fashion the anti-tumor activity of the combination of Alemtuzumab and EPOCH chemotherapy.

Eligibility:

CD52-expressing lymphoid malignancy.

Patients with chemotherapy naive aggressive T & NK lymphomas. Patients with alk-positive anaplastic large cell lymphoma and patients with T cell precursor disease are not eligible.

Age greater than or equal to 17 years.

Adequate organ function, unless impairment due to respective organ involvement by tumor.

No active symptomatic ischemic heart disease, myocardial infarction or congestive heart. failure within the past year.

Human immunodeficiency virus (HIV) negative.

Not pregnant or nursing.

Design:

Three dose levels of Alemtuzumab will be evaluated to determine the toxicity profile and in a preliminary fashion the antitumor activity of the combination with Dose-Adjusted EPOCH.

Three dose levels of Alemtuzumab will be explored, in cohorts of three to six patients each. Patients will receive either 30, 60, or 90 mg of Alemtuzumab on day 1 of therapy, followed by dose-adjusted EPOCH chemotherapy days 1-5.

DETAILED DESCRIPTION:
Background:

The paradigm of combining therapeutic agents with non-overlapping toxicities for the treatment of malignancy produces clinical remissions and cures in a number of tumor types.

A new class of agents, humanized and chimerized monoclonal antibodies, typically have little or no hematopoietic toxicity and can be readily combined with full doses of cytotoxic chemotherapy. It has become clear that in certain lymphomas and breast cancers, the combination of monoclonal antibodies and chemotherapy improves response rate and the quality of the response compared with that achieved by treatment with either agent alone.

The clinical outcome for patients with T-cell non-Hodgkins lymphoma is significantly inferior to the outcome of patients with B-cell non-Hodgkins lymphoma. In most reports less than 20% of patients with T cell lymphoid malignancies remain free of disease at 5 years.

Objective:

Determine the toxicity and maximum tolerated dose (MTD) of Alemtuzumab and EPOCH chemotherapy in untreated cluster of differentiation 52 (CD52)-expressing T and natural killer (NK) lymphoid malignancies

Eligibility:

* CD52-expressing lymphoid malignancy.
* Patients with chemotherapy naive aggressive T & NK lymphomas. Patients with alk-positive anaplastic large cell lymphoma and patients with T cell precursor disease are not eligible.
* Age greater than or equal to 17 years.
* Adequate organ function, unless impairment due to respective organ involvement by tumor.
* No active symptomatic ischemic heart disease, myocardial infarction or congestive heart. failure within the past year.
* Human immunodeficiency virus (HIV) negative.
* Not pregnant or nursing.

Design:

Three dose levels of Alemtuzumab will be evaluated to determine the toxicity profile and in a preliminary fashion the antitumor activity of the combination with Dose-Adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH).

Three dose levels of Alemtuzumab will be explored, in cohorts of three to six patients each. Patients will receive either 30, 60, or 90 mg of Alemtuzumab on day 1 of therapy, followed by dose-adjusted EPOCH chemotherapy days 1-5.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Cluster of differentiation 52 (CD52)-expressing lymphoid malignancy, confirmed by pathology or flow cytometry staff of the Hematopathology Section, Laboratory of Pathology, National Cancer Institute (NCI). Patients with T & natural killer (NK) cell malignancy without accessible tissue for flow cytometry analysis may be treated on this study.

Patients with chemotherapy naive aggressive T & NK lymphomas, including but not limited to peripheral T cell lymphoma (not otherwise specified (nos)), gamma-delta hepatosplenic T cell lymphoma, subcutaneous panniculitis-like T cell, NK-T cell lymphoma confirmed by pathology or flow cytometry staff of the Hematopathology Section, Laboratory of Pathology, NCI. Patients with alk-positive anaplastic large cell lymphoma and patients with T cell precursor disease are not eligible.

Age greater than or equal to 17 years.

Laboratory tests: Creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than or equal to 60 ml/min; bilirubin less than 2.0 mg/dl unless due to Gilbert's, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 times upper limit of normal (ULN) (AST and ALT is less than or equal to 6 times ULN for patients on hyperalimentation for whom these abnormalities are felt to be due to the hyperalimentation) and; absolute neutrophil count (ANC) is greater than or equal to 1000/mm(3), platelet greater than or equal to 75,000/mm(3); unless impairment due to respective organ involvement by tumor.

No active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year.

Human immunodeficiency virus (HIV) negative, because of the unknown effects of combined therapy with chemotherapy and an immunosuppressive agent on HIV progression.

Signed informed consent.

Willing to use contraception.

Not pregnant or nursing, because of the unknown effects of Alemtuzumab on the developing fetus and infant.

No serious underlying medical condition or infection that would contraindicate treatment. Patients with central nervous system (CNS) involvement are eligible for treatment on this study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-09-19 (Actual); Primary Completion 2009-06-11 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wing MG, Moreau T, Greenwood J, Smith RM, Hale G, Isaacs J, Waldmann H, Lachmann PJ, Compston A. Mechanism of first-dose cytokine-release syndrome by CAMPATH 1-H: involvement of CD16 (FcgammaRIII) and CD11a/CD18 (LFA-1) on NK cells. J Clin Invest. 1996 Dec 15;98(12):2819-26. doi: 10.1172/JCI119110. PMID 8981930
- [Background] Harris NL, Jaffe ES, Stein H, Banks PM, Chan JK, Cleary ML, Delsol G, De Wolf-Peeters C, Falini B, Gatter KC, et al. A revised European-American classification of lymphoid neoplasms: a proposal from the International Lymphoma Study Group. Blood. 1994 Sep 1;84(5):1361-92. No abstract available. PMID 8068936
- [Background] A clinical evaluation of the International Lymphoma Study Group classification of non-Hodgkin's lymphoma. The Non-Hodgkin's Lymphoma Classification Project. Blood. 1997 Jun 1;89(11):3909-18. PMID 9166827
- [Derived] Lai C, Cole DE, Steinberg SM, Lucas N, Dombi E, Melani C, Roschewski M, Balis F, Widemann BC, Wilson WH. Doxorubicin pharmacokinetics and toxicity in patients with aggressive lymphoma and hepatic impairment. Blood Adv. 2023 Feb 28;7(4):529-532. doi: 10.1182/bloodadvances.2022007431. PMID 35882475
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-C-0304.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Alemtuzumab 30 mg: Alemtuzumab (Campath) 30mg intravenous (IV) on day 1 of therapy, followed by etoposide (50mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), prednisone (60mg/m(2) day by mouth (PO) day 0-5), vincristine (0.4mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), cyclophosphamide (750mg/m(2) day intravenous day 5), doxorubicin (10mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), (EPOCH) days 1-5 every 3 weeks for up to 6 cycles.
- Alemtuzumab 60 mg: Alemtuzumab (Campath) 60mg intravenous (IV) on day 1 of therapy, followed by etoposide (50mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), prednisone (60mg/m(2) day by mouth (PO) day 0-5), vincristine (0.4mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), cyclophosphamide (750mg/m(2) day intravenous day 5), doxorubicin (10mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), (EPOCH) days 1-5 every 3 weeks for up to 6 cycles.
- Alemtuzumab 90 mg: Alemtuzumab (Campath) 90mg intravenous (IV) on day 1 of therapy, followed by etoposide (50mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), prednisone (60mg/m(2) day by mouth (PO) day 0-5), vincristine (0.4mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), cyclophosphamide (750mg/m(2) day intravenous day 5), doxorubicin (10mg/m(2) day continuous intravenous (CIV) day 1-4 (96 hours)), (EPOCH) days 1-5 every 3 weeks for up to 6 cycles.
Period: Cohort 1 - Dose Level 1 (Weeks 1 - 18)
Arm/Group | Alemtuzumab 30 mg | Alemtuzumab 60 mg | Alemtuzumab 90 mg
Started | 25 | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 9 | 0 | 0
Not completed — Toxicity | 9 | 0 | 0
Period: Cohort 2 - Dose Level 2 (Weeks 1-18)
Arm/Group | Alemtuzumab 30 mg | Alemtuzumab 60 mg | Alemtuzumab 90 mg
Started | 0 | 3 | 0
Completed | 0 | 1 | 0
Not Completed | 0 | 2 | 0
Not completed — Toxicity | 0 | 2 | 0
Period: Cohort 3 - Dose Level 3 (Weeks 1-18)
Arm/Group | Alemtuzumab 30 mg | Alemtuzumab 60 mg | Alemtuzumab 90 mg
Started | 0 | 0 | 3
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 2
Not completed — Toxicity | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received at least one dose of Alemtuzumab (Campath) 30mg, 60mg, or 90mg on day 1 of therapy followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) chemotherapy intravenously every 3 weeks for up to 6 cycles.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 27
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.52 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Alemtuzumab
Description: MTD was achieved by increasing doses of Alemtuzumab on three cohorts. Cohort 1 received 30mg of Alemtuzumab, cohort 2 received 60mg of Alemtuzumab, and cohort 3 received 90mg of Alemtuzumab intravenously up to 2 cycles. The MTD reflects the highest dose of Alemtuzumab in which no more than 1 of 6 participants entered at a specific dose level experienced a dose limiting toxicity (DLT).
Time Frame: up to 2 cycles of therapy, approximately 42 days
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 31
mg | 30

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 67 months and 9 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
Participants | 31

3. Secondary Outcome: Clinical Response
Description: Response was measured by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas. Complete remission (CR) is complete disappearance of all detectable clinical and radiographic evidence of disease. Complete response unconfirmed (Cru)is as per complete remission criterion except that if a residual node is greater than 1.5cm, it must have decreased by greater than 75% in the sum of the products of the perpendicular diameters (SPD). Partial response (PR) is ≥50% decrease in the SPD of 6 largest dominant nodes or nodal masses. Progressive disease (PD) is ≥50% increase from the nadir in the SPD of any previously identified abnormal node for PRS or non-responders. Stable disease (SD) is less than a PR but not progressive disease.
Time Frame: From date of onstudy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 67 months and 9 days.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who received at least one dose of Alemtuzumab (Campath) 30mg, 60mg, or 90mg on day 1 of therapy followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) chemotherapy intravenously every 3 weeks for up to 6 cycles.
  The adverse events are not reported per dose level because we normally look at all adverse events together irrespective of the dose level.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Participants
  Complete Response | 17
  Complete Response Unconfirmed | 0
  Partial Response | 7
  Progressive Disease | 2
  Stable Disease | 1
  Not Evaluable | 4

ADVERSE EVENTS:
Time Frame: 67 months and 9 days
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 23/31
Serious Adverse Events (participants affected / at risk) | 23/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=31)
DEATH:: Death related to the study (General disorders) | 7 (7)
DEATH:: Death due to progression (General disorders) | 16 (16)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Upper GI Not otherwise specified (NOS) (Blood and lymphatic system disorders) | 1 (1)
INFECTION:: Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
INFECTION:: Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Blood
INFECTION:: Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Brain (encephalitis, infectious)
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) — (ANC <1.0 x 10e9/L):: Lung (pneumonia)
INFECTION:: Infection with unknown ANC:: Blood (Infections and infestations) | 1 (1)
RENAL/GENITOURINARY:: Cystitis (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY:: Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=31)
ALLERGY/IMMUNOLOGY:: Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 7 (11)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 9 (11)
AUDITORY/EAR:: Otitis, middle ear (non-infectious) (Blood and lymphatic system disorders) | 1 (1)
AUDITORY/EAR:: Tinnitus (Ear and labyrinth disorders) | 1 (1)
BLOOD/BONE MARROW:: Bone marrow cellularity (Blood and lymphatic system disorders) | 4 (4)
BLOOD/BONE MARROW:: Hemoglobin (Blood and lymphatic system disorders) | 29 (101)
BLOOD/BONE MARROW:: Leukocytes (total white blood count (WBC)) (Blood and lymphatic system disorders) | 30 (121)
BLOOD/BONE MARROW:: Lymphopenia (Blood and lymphatic system disorders) | 30 (74)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 30 (116) — Absolute neutrophil count/absolute granulocyte count (ANC/AGC)
BLOOD/BONE MARROW:: Platelets (Cardiac disorders) | 28 (102)
CARDIAC ARRHYTHMIA:: Palpitations (Cardiac disorders) | 2 (2)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus bradycardia (Blood and lymphatic system disorders) | 1 (1)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus tachycardia (Cardiac disorders) | 1 (1)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Supraventricular arrhythmia NOS (General disorders) | 1 (1) — Not otherwise specified (NOS)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Supraventricular tachycardia (General disorders) | 2 (2)
CARDIAC ARRHYTHMIA:: Vasovagal episode (Cardiac disorders) | 1 (1)
CARDIAC GENERAL:: Hypertension (Cardiac disorders) | 1 (1)
CARDIAC GENERAL:: Hypotension (Cardiac disorders) | 9 (14)
COAGULATION:: PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 4 (5)
CONSTITUTIONAL SYMPTOMS:: Fatigue (asthenia, lethargy, malaise) (General disorders) | 18 (33)
CONSTITUTIONAL SYMPTOMS (General disorders) | 11 (16) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
CONSTITUTIONAL SYMPTOMS:: Insomnia (General disorders) | 5 (5)
CONSTITUTIONAL SYMPTOMS:: Rigors/chills (General disorders) | 9 (14)
CONSTITUTIONAL SYMPTOMS:: Sweating (diaphoresis) (General disorders) | 4 (4)
CONSTITUTIONAL SYMPTOMS:: Weight loss (General disorders) | 7 (8)
DERMATOLOGY/SKIN:: Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin - Other (Specify, excoriation) (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 15 (15)
DERMATOLOGY/SKIN:: Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
DERMATOLOGY/SKIN:: Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Nail changes (Skin and subcutaneous tissue disorders) | 5 (5)
DERMATOLOGY/SKIN:: Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (4)
DERMATOLOGY/SKIN:: Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (12)
DERMATOLOGY/SKIN:: Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 11 (15)
GASTROINTESTINAL:: Constipation (Gastrointestinal disorders) | 12 (14)
GASTROINTESTINAL:: Dehydration (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Dental: teeth (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Diarrhea (Gastrointestinal disorders) | 14 (23)
GASTROINTESTINAL:: Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL:: Esophagitis (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Flatulence (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL:: Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Specify, duodenitis) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4)
GASTROINTESTINAL:: Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Mucositis/stomatitis (clinical exam):: Oral cavity (Gastrointestinal disorders) | 20 (33)
GASTROINTESTINAL:: Mucositis/stomatitis (clinical exam):: Pharynx (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Mucositis/stomatitis (functional/symptomatic):: Esophagus (Blood and lymphatic system disorders) | 1 (1)
GASTROINTESTINAL:: Mucositis/stomatitis (functional/symptomatic):: Oral cavity (Gastrointestinal disorders) | 7 (8)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 18 (38)
GASTROINTESTINAL:: Proctitis (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4 (4)
GASTROINTESTINAL:: Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 13 (20)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Lower GI NOS (Gastrointestinal disorders) | 1 (1) — Not otherwise specified (NOS)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Oral cavity (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Upper GI NOS (Gastrointestinal disorders) | 2 (2)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Bladder (Renal and urinary disorders) | 1 (1) — Genitourinary (GU)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Urinary NOS (Renal and urinary disorders) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage, pulmonary/upper respiratory:: Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage, pulmonary/upper respiratory:: Nose (Metabolism and nutrition disorders) | 4 (5)
HEMORRHAGE/BLEEDING:: Hemorrhage/Bleeding - Other (Specify, R. neck after picc line) (General disorders) | 1 (1)
HEMORRHAGE/BLEEDING:: Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
INFECTION:: Febrile neutropenia (Metabolism and nutrition disorders) | 16 (28) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
INFECTION:: Infection(documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) — (ANC <1.0 x 10e9/L):: Abdomen NOS
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (2) — (ANC <1.0 x 10e9/L):: Bladder (urinary)
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 4 (5) — (ANC <1.0 x 10e9/L):: Blood
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (2) — (ANC <1.0 x 10e9/L):: Brain (encephalitis, infectious)
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Nervous system disorders) | 1 (1) — (ANC <1.0 x 10e9/L):: Catheter-related
INFECTION:Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Nervous system disorders) | 1 (1) — (ANC <1.0 x 10e9/L):: Cecum
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Nervous system disorders) | 1 (1) — (ANC <1.0 x 10e9/L):: Colon
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Nervous system disorders) | 1 (1) — (ANC <1.0 x 10e9/L):: Conjunctiva
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Nervous system disorders) | 1 (1) — (ANC <1.0 x 10e9/L):: Lung (pneumonia)
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (2) — (ANC <1.0 x 10e9/L):: Mucosa
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) — (ANC <1.0 x 10e9/L):: Spleen
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 4 (4) — (Absolute neutrophil count (ANC) <1.0 x 10e9/L):: Urinary tract NOS
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (5) — (ANC <1.0 x 10e9/L):: Vein
INFECTION:: Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Musculoskeletal and connective tissue disorders) | 2 (2) — (ANC <1.0 x 10e9/L):: Wound
INFECTION:: Infection - Other (Specify, BLOOD) (Gastrointestinal disorders) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Blood (Infections and infestations) | 1 (3)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Sinus (Musculoskeletal and connective tissue disorders) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Skin (cellulitis) (Infections and infestations) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Urinary tract NOS (Infections and infestations) | 4 (4) — Not otherwise specified (NOS)
INFECTION:: Infection with unknown ANC:: Blood (Musculoskeletal and connective tissue disorders) | 1 (1)
INFECTION:: Infection with unknown ANC:: Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
INFECTION:: Infection with unknown ANC:: Urinary tract NOS (Infections and infestations) | 1 (1)
LYMPHATICS:: Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
LYMPHATICS:: Edema: limb (Blood and lymphatic system disorders) | 4 (4)
LYMPHATICS:: Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
METABOLIC/LABORATORY:: ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 14 (38) — alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT)
METABOLIC/LABORATORY:: AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 14 (29) — aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT)
METABOLIC/LABORATORY:: Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 20 (49)
METABOLIC/LABORATORY:: Alkaline phosphatase (Metabolism and nutrition disorders) | 16 (22)
METABOLIC/LABORATORY:: Amylase (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Bicarbonate, serum-low (Metabolism and nutrition disorders) | 4 (6)
METABOLIC/LABORATORY:: Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 10 (12)
METABOLIC/LABORATORY:: Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
METABOLIC/LABORATORY:: Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 19 (44)
METABOLIC/LABORATORY:: Creatinine (Metabolism and nutrition disorders) | 3 (3)
METABOLIC/LABORATORY:: Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 17 (47)
METABOLIC/LABORATORY:: Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 (6)
METABOLIC/LABORATORY:: Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 15 (30)
METABOLIC/LABORATORY:: Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 18 (28)
METABOLIC/LABORATORY:: Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 16 (26)
METABOLIC/LABORATORY:: Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 9 (10)
METABOLIC/LABORATORY:: Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 17 (26)
METABOLIC/LABORATORY:: Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 4 (4)
METABOLIC/LABORATORY:: Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 16 (28)
METABOLIC/LABORATORY:: Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (5)
MUSCULOSKELETAL/SOFT TISSUE:: Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE:: Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE:: Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) — Extremity-lower
MUSCULOSKELETAL/SOFT TISSUE:: Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) — Whole body/generalized
MUSCULOSKELETAL/SOFT TISSUE:: Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1) — cervical spine range of motion
MUSCULOSKELETAL/SOFT TISSUE:: Soft tissue necrosis:: Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUROLOGY:: Confusion (Nervous system disorders) | 3 (3)
NEUROLOGY:: Dizziness (Nervous system disorders) | 9 (12)
NEUROLOGY:: Laryngeal nerve dysfunction (Nervous system disorders) | 1 (1)
NEUROLOGY:: Mood alteration:: Agitation (Nervous system disorders) | 1 (1)
NEUROLOGY:: Mood alteration:: Anxiety (Nervous system disorders) | 3 (3)
NEUROLOGY:: Mood alteration:: Depression (Nervous system disorders) | 1 (1)
NEUROLOGY:: Neuropathy: motor (Nervous system disorders) | 3 (3)
NEUROLOGY:: Neuropathy: sensory (Nervous system disorders) | 24 (24)
NEUROLOGY:: Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
NEUROLOGY:: Syncope (fainting) (Nervous system disorders) | 2 (2)
NEUROLOGY:: Tremor (Nervous system disorders) | 1 (1)
OCULAR/VISUAL:: Ocular/Visual - Other (Specify, red eyes) (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Vision-blurred vision (Eye disorders) | 3 (3)
OCULAR/VISUAL:: Vision-photophobia (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
PAIN:: Pain - Other (Specify, L wrist) (General disorders) | 1 (1)
PAIN:: Pain:: Abdomen Not otherwise specified (NOS) (Gastrointestinal disorders) | 7 (9)
PAIN:: Pain:: Back (Musculoskeletal and connective tissue disorders) | 7 (9)
PAIN:: Pain:: Bladder (Renal and urinary disorders) | 1 (1)
PAIN:: Pain:: Bone (Musculoskeletal and connective tissue disorders) | 12 (20)
PAIN:: Pain:: Buttock (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain:: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 5 (6)
PAIN:: Pain:: Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
PAIN:: Pain:: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain:: Eye (Eye disorders) | 2 (2)
PAIN:: Pain:: Head/headache (Nervous system disorders) | 13 (22)
PAIN:: Pain:: Joint (Musculoskeletal and connective tissue disorders) | 5 (6)
PAIN:: Pain:: Muscle (Musculoskeletal and connective tissue disorders) | 10 (11)
PAIN:: Pain:: Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain:: Rectum (Gastrointestinal disorders) | 1 (1)
PAIN:: Pain:: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PULMONARY/UPPER RESPIRATORY:: Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
PULMONARY/UPPER RESPIRATORY:: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (8)
PULMONARY/UPPER RESPIRATORY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY/UPPER RESPIRATORY:: Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
PULMONARY/UPPER RESPIRATORY:: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL/GENITOURINARY:: Cystitis (Renal and urinary disorders) | 6 (6)
RENAL/GENITOURINARY:: Incontinence, urinary (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY:: Obstruction, GU:: Ureter (Renal and urinary disorders) | 1 (1) — Genitourinary (GU)
RENAL/GENITOURINARY:: Urinary frequency/urgency (Renal and urinary disorders) | 5 (6)
VASCULAR:: Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
VASCULAR:: Thrombosis/embolism (vascular access-related) (Vascular disorders) | 3 (3)
VASCULAR:: Thrombosis/thrombus/embolism (Vascular disorders) | 5 (5)
GASTROINTESTINAL:: Gastrointestinal - Other (Specify, tongue-blue spot) (Gastrointestinal disorders) | 1 (1)
OCULAR/VISUAL:: Ocular/Visual - Other (Specify, dilated, non-reactive R.pupil (Eye disorders) | 1 (1)
PAIN:: Pain - Other (Specify, lumbar puncture (LP) site) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain - Other (Specify, Pain L big toe (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain - Other (Specify, Pain: jaw pain) (Gastrointestinal disorders) | 1 (1)
PAIN:: Pain - Other (Specify, Pain:teeth) (Gastrointestinal disorders) | 1 (2)
PAIN:: Pain - Other (Specify, Pain: tooth (Gastrointestinal disorders) | 1 (1)
PAIN:: Pain - Other (Specify, Pain:groin) (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT00069238/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT00069238/ICF_002.pdf